CLINICAL TRIAL: NCT06857981
Title: Patient's Database: Prepare for Your Surgery Program
Status: Recruiting | Type: Observational
Sponsor: Pontificia Universidad Catolica de Chile (Other)
Responsible Party: Sponsor
Other Study IDs: 241120002; 241120002 (Other Grant/Funding Number: P100 Red Salud UC Christus)
Record Dates: First submitted 2025-02-24; First posted 2025-03-05 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: Frailty in Adult Surgery; Frail Elderly Syndrome; Database; Perioperative Care; Prehabilitation
Keywords: Database; Perioperative care; Prospective Studies; Frailty; Follow-Up Studies; Prehabilitation
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient's Data Base: Patients referred to the Prepare for Your Surgery program
  Interventions: Other: Clinical data collection

INTERVENTIONS:
Other: Clinical data collection — Patient's data will be collected, including: date of birth, age, gender/sex, pathology for admission, comorbidities, treatment received, and proposed interventions based on initial assessment.

SUMMARY:
Frailty is a multidimensional syndrome that predominantly affects older people and people with long-term treatments such as cancer and chronic pain. This results in an increased risk of disability, reduced resistance and greater vulnerability to stressors.

These factors culminate in worse postoperative outcomes, including higher rates of complications and mortality. With the current demographic shift towards an aging population in Latin America and Chile, the prevalence of frailty among surgical patients is increasing.

Despite the clear association between frailty and adverse postoperative effects, in Chile there are few centers that routinely perform objective preoperative frailty assessment before to surgery. This is due to logistical challenges, the need for specialized training, and assessment tools. As a result, frailty remains an underestimated syndrome in the perioperative setting.

Various interventions have been proposed to improve the care of fragile surgical patients. Prehabilitation, a multidisciplinary program designed to prepare patients for surgery and improve their resilience to surgical stress, has emerged as a promising intervention. Recent studies indicate that prehabilitation may lead to shorter hospital length of stay (LOS) and fewer complications.

Recognizing the vital role that frailty plays in surgical outcomes and the paucity of research on prehabilitation, a prehabilitation or timely presurgical conditioning program (Prepare for Your Surgery Program) has been implemented at our center. This proposal seeks to optimize the patient before a surgical intervention in order to reduce frailty and complications, thus improving recovery and medium-term results.

The program consists of interventions 4 to 6 weeks before surgery focused on: nursing assessment, screening and follow-up, geriatric and/or internal medicine assessment and intervention, physiotherapy assessment and intervention, nutrition assessment and intervention, psychological assessment and intervention, and preoperative anesthesiology intervention.

For this purpose, it has been proposed to create a prospective database of patients from the Prepare for Your Surgery Program, who undergo elective surgery at Hospital Clinico Red Salud UC-Christus.

DETAILED DESCRIPTION:
Potential participants in the "Prepare for Your Surgery" program must complete the informed consent process, having met the inclusion criteria for this database. Demographic data will be collected from patients, including: date of birth, age, gender/sex, pathology for which they were admitted, comorbidities, treatment they receive, and proposed interventions according to their initial evaluation. In turn, the episode number will be stored, whether their pathology is covered by the public health system through Explicit Health Guarantees (GES) or not, the number of days hospitalized associated with the surgical episode, specialty to which it corresponds, and the type of surgery according to code. From the clinical part, the data from your medical record will be stored, specifically, the results of the application of the following tests and index calculations.

Regarding the program, it consists mainly of 7 stages:

1. An evaluation by the nurse navigator who will carry out the screenings defined by the treating team (in person or online). The instruments to be applied consist of the evaluation of frailty (Clinical Frailty Scale CFS, FRAIL Scale, FRIED phenotype); cognitive assessment using the Montreal Cognitive Assessment (MoCA) or Mini Cog; functionality (Barthel Index); Revised Cardiovascular Risk Index (Lee); Charlson Comorbidity Index nicotine dependence (Fageström Test); evaluation of obstructive sleep apnea (STOP Bang); stroke risk scale (CHAD VASc2); Respiratory failure index (Arozullah Respiratory Failure Index); Hospital Anxiety and Depression Scale (PHQ-2); evaluation of nutritional status (Mini Nutritional Assessment MNA); pain assessment (PROMIS pain); Physical Functioning Assessment (PROMIS PF), 6-Minute Walking Test, Grip Strength (Handgrip Test) and the Short Physical Performance Test (SPPT).
2. A 30-minute outpatient medical consultation will be carried out that will focus on the evaluation and optimization of comorbidities, pre-surgical indications, request for examinations, referral to specialists, among others (in-person).
3. 8 to 10 kinesiology evaluation and intervention sessions will be carried out according to the physical-functional status of the patient.
4. 1 to 2 nutritional interventions will be carried out on physical-functional nutritional-metabolic status.
5. If necessary, contact via email, telephone and/or telematics or with the results of the examinations will be used and define if a second consultation is justified, coordinated with the nurse navigator.
6. Intra-hospital indicators will be recorded and monitored: days of hospitalization (surgical complications according to the Clavien Dindo classification or surgical risk indexes), daily in-hospital destination (basic care room, intermediate care room and/or ICU), until discharge.
7. Post-hospital discharge follow-up will be carried out on complications, readmissions, mortality and/or relevant history of the patients for 3 to 6 months according to the surgical specialty.

The data to be obtained are clinically recorded and will be stored in the TrakCare program's own databases in the electronic record systems of the Hospital Clinico Red UC-CHRISTUS, surgical table (SAQ), SAP and other related systems. For data extraction, an encrypted data table associated with the "episode" numbering generated sequentially by the SAP care systems has been proposed. Each access to the "Patient Database: Prepare for Your Surgery Program" will be restricted by the team responsible for the database, which is accessed by means of a username and password with encrypted restrictions on the data generated.

To guarantee the confidentiality of the data, alternate identifiers will be used (example Male = 1, Female =2), which are codes associated with a case, which can bring together several episodes, to which numbers and letters are assigned, for which They are considered encrypted data without sensitive data. The encoded data can only be accessed by the responsible team who will guarantee the internal traceability of the data, safeguarding confidentiality and providing anonymized and/or encoded forms of the data collected. In addition, the data is kept linked to the clinical record servers which have their own backup and security systems within the services provided to the Hospital Clinico Red UC-CHRISTUS.

Once the number of participants is complete, the recorded data will be analyzed to describe the characteristics of the patients included in this type of program, evaluate key indicators such as adherence, participation and in the future generate improvements in implementation protocols, national or local policies and generate publications related to this topic.

ELIGIBILITY:
Inclusion Criteria:

* Patients referred to the Prepare for Your Surgery program
* Patients characterized as frail according to the Clinical Frailty Scale (score ≥ 4), FRAIL scale or FRIED frailty phenotype or the clinical judgment of the referring surgeon, with at least 4 weeks to receive surgery
* Elective surgery to be performed at Hospital Clinico Red de Salud UC-Christus

Exclusion Criteria:

* Patients who will not undergo elective surgery at Hospital Clínico Red de Salud UC-Christus.
* Patients who require emergency surgery
* Patients who for various reasons cannot comply with the interventions proposed for this preparation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are users of the Hospital Clinico Red de Salud UC-Christus who are going to undergo elective surgery to be performed at the same center
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2025-05-21 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Establishment of a database | 1 month
  Establish a database to record the demographic characteristics, frailty and/or comorbidities and relevant preoperative history of patients referred to the "Prepare for your Surgery" program.

SECONDARY OUTCOMES:
Registry of in-hospital history | 1 month
  Record surgical, anesthetic, hospital stay and/or relevant in-hospital history of patients admitted to the "Prepare for Your Surgery" program.
Patient Follow-Up | 3 - 6 months
  Record the characteristics of possible complications, rehospitalizations, mortality, and/or relevant histories of patients 3 to 6 months after hospital discharge, according to their surgical specialty.

CONTACTS AND LOCATIONS:
Overall Officials: Victor Contreras, MSN, Principal Investigator — Pontificia Universidad Catolica de Chile
Locations (2):
- Chile (2):
  - Pontificia Universidad Católica de Chile, Santiago, Santiago Metropolitan
  - Red de Salud UC Christus, Santiago

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gibbison B, Pufulete M. Prehabilitation before cardiac surgery. Br J Anaesth. 2025 Jan;134(1):5-7. doi: 10.1016/j.bja.2024.11.001. Epub 2024 Nov 26. PMID 39603851
- [Background] Gillis C, Ljungqvist O, Carli F. Prehabilitation, enhanced recovery after surgery, or both? A narrative review. Br J Anaesth. 2022 Mar;128(3):434-448. doi: 10.1016/j.bja.2021.12.007. Epub 2022 Jan 7. PMID 35012741
- [Background] Contreras V, Elgueta MF, Balde D, Astaburuaga P, Carrasco M, Pedemonte JC, Nicoletti MN, Medina Diaz R, Franco S, Agurto R, Vivanco C, Figueroa C, Alamos M, Cuzmar Benitez V, Vargas B, Barraza B, Rematal C, Cortinez LI. Prehabilitation for Chilean frail elderly people - pre-surgical conditioning protocol - to reduce the length of stay: randomized control trial. Minerva Anestesiol. 2024 Dec;90(12):1098-1107. doi: 10.23736/S0375-9393.24.18245-4. PMID 39836361